CLINICAL TRIAL: NCT04911517
Title: Rationale and Design of a Prospective, Multicenter Phase Ⅱ Clinical Trial of Safety and Efficacy Evaluation of Long Course Neoadjuvant Chemoradiotherapy Plus Tislelizumab Followed by TME for LARC.
Brief Title: Neoadjuvant Chemoradiotherapy Plus Tislelizumab Followed by TME for LARC.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Friendship Hospital (Other)
Collaborators: Hangzhou New Horizon Health Technology Co., Ltd. (Unknown); BeOne Medicines (Industry); Beijing Chao Yang Hospital (Other); Xuanwu Hospital, Beijing (Other); Tianjin Medical University General Hospital (Other); People's Hospital of Tianjin (Unknown); Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Principal Investigator, Zhongtao Zhang, professor, Beijing Friendship Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BFH-NCRTPD
Record Dates: First submitted 2021-05-23; First posted 2021-06-03 (Actual); Last update posted 2022-02-23 (Actual); Status verified 2022-02

CONDITIONS: Colorectal Neoplasms
Keywords: Colorectal Neoplasms; Programmed Cell Death 1 Receptor; Neoadjuvant Therapy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Capecitabine

STUDY DESIGN:
Intervention Model Description: The enrolled patients in this NCRT-PD-1-LARC trial will receive long course radiotherapy (50 Gy/25 f, 2 Gy/f, 5 days/week) and three 21-day cycles capecitabine (1000 mg/m2, bid, po, day1-14) plus three 21-day cycles tislelizumab (200 mg, iv.gtt, day8), followed by total mesorecta excision 6-8 week after the end of radiotherapy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- long course radiotherapy + capecitabine + PD-1 monoclonal antibody treatment combinations (Experimental): long course radiotherapy + capecitabine + PD-1 monoclonal antibody treatment combinations in patients with locally advanced rectal cancer
  Interventions: Combination Product: long course radiotherapy + capecitabine + PD-1 monoclonal antibody treatment combinations

INTERVENTIONS:
Combination Product: long course radiotherapy + capecitabine + PD-1 monoclonal antibody treatment combinations — long course radiotherapy + capecitabine + PD-1 monoclonal antibody treatment combinations in patients with locally advanced rectal cancer

SUMMARY:
Long course radiotherapy plus neoadjuvant chemotherapy followed by resection total mesorecta excision has accepted widespread recognized in the treatment of locally advanced rectal cancer (LARC). Tislelizumab, an anti-PD1(programmed death 1) humanized IgG4 (Immunoglomin G4) monoclonal antibody, has been demonstrated with clinical activity and is approved for treating recurrent/refractory classical Hodgkin lymphoma and locally advanced/metastatic urothelial carcinoma in China.

The aim of This NCRT-PD-1-LARC trial is to evaluate the efficacy and safety of long course neoadjuvant chemoradiotherapy plus tislelizumab followed by total mesorecta excision for LARC. This NCRT-PD-1-LARC trial will be a prospective, multicenter and phase Ⅱ clinical trial designed to evaluate the safety and efficacy of LARC patients treated with long course neoadjuvant chemoradiotherapy plus tislelizumab followed by total mesorecta excision. It will consecutively enroll 50 stage II/III LARC patients (cT3N0M0 and cT1-3N1-2M0) with the tumor distal location ≤ 10cm from anal verge at 7 centers in China. The enrolled patients will receive long course radiotherapy (50 Gy/25 f, 2 Gy/f, 5 days/week) and three 21-day cycles capecitabine (1000 mg/m2, bid, po, day1-14) plus three 21-day cycles tislelizumab (200 mg, iv.gtt, day8), followed by total mesorecta excision 6-12 week after the end of radiotherapy. The primary efficacy endpoint will be the pathological complete response (pCR) rate, which is defined as absence of viable tumor cells in the primary tumor and lymph nodes.

ELIGIBILITY:
Inclusion criteria:

* Patients have been fully aware of the content of this study and signed the informed consent voluntarily;
* Patients with rectal cancers must satisfied all the following conditions: Stage II/III LARC (cT1-3N1-2M0)；Tumor distal location ≤10 cm from anal verge (MRI diagnosed);
* Patients regardless of gender with aged ≥18 years and ECOG score of 0 or 1;
* Physical and viscera function of patients can withstand major abdominal surgery;
* Patients are willing and able to follow the study protocol during the study;
* Patients give consent to the use of blood and pathological specimens for study;
* Within 28 days prior to enrolment, we must confirm a negative serological pregnancy test for child-bearing age women and they agree to use effective contraception for the duration of drug use and for 60 days after the last dose.

Exclusion criteria:

* Patients have a present or previous active malignancy except the diagnosis of rectal cancer this time;
* Patients underwent major surgery within 4 weeks prior to study treatment;
* Patients have any condition affects the absorption of capecitabine through gastrointestinal tract;
* Patients have severe uncontrolled recurrent infections, or other severe uncontrolled concomitant diseases;
* Patients who are allergic to any of the ingredients under study;
* Patients with severe concomitant diseases with estimated survival ≤ 5 years;
* Patients with present or previous moderate or severe liver and kidney damage presently or previously;
* Patients have received other study medications or any immunotherapy currently or in the past;
* Patients preparing for or previously received organ or bone marrow transplant;
* Patients who received immunosuppressive or systemic hormone therapy for immunosuppressive purposes within 1 month prior to the initiation of study therapy;
* Patients with congenital or acquired immune deficiency (such as HIV infection);
* If patients with a history of uncontrolled epilepsy, central nervous system disease or mental disorder, the investigator will determine whether the clinical severity prevents the signing of informed consent or affects the patient's oral medication compliance;
* Patients with other factors that may affect the study results or cause the study to be terminated midway, such as alcoholism, drug abuse, other serious diseases (including mental illness) requiring combined treatment and severe laboratory examination abnormalities.
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
pathologic complete response（pCR） | 1 year
  All the enrolled patients will receive total mesorectal excision (TME) 7-9 weeks after the end of long course radiotherapy. The rectal specimens will be evaluated by the pathologists who are experienced on the rectal cancer diagnosis according to the 1997 Dworak grading system. The rectal cancer will be classified into 5 grades. Grade 0-3 will be considered as non-pCR while grade 4 represent pCR.

SECONDARY OUTCOMES:
neoadjuvant rectal (NAR) score | 1 year
  The neoadjuvant rectal (NAR) score is a promising indicator of survival after preoperative chemoradiotherapy for rectal cancer. The NAR score was calculated according to the following formula: NAR score = [5pN - 3(cT - pT) + 12]2∕9.61. (clinical tumor (cT) stage, pathologic tumor (pT) stage, pathologic nodal (pN) stage)
objective response rate (ORR) | 1 year
  ORR is evaluated according to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1. The ORR rate is the sum of complete response (CR) and partial response (PR)
R0 resection rate | 1 year
  During the surgical process, the surgeon will evaluate the level of cancer resection. It will be classified as R0, R1, R2 resection. Therefore, we can calculate R0 resection rate.
anal preservation rate | 1 year
  the surgeon will decide whether the anal can be preserved on the basis of the rectal cancer and intraoperative situation. anal preservation rate is the percentage of patients who achieve anal preservation.
3-year local recurrence rate (LRR) | 3 year
  During the 3-year follow-up, the percentage of local recurrence.
3-year disease free survival (DFS) | 3 year
  During the 3-year follow-up, the percentage of the patients who is disease free.
3-year overall survival (OS) | 3 year
  During the 3-year follow-up, the percentage of the patients who is sill survival at the end of follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: yaohongwei@ccmu.edu.cn Yao, Dr., Study Chair — Department of General Surgery, Beijing Friendship Hospital, Capital Medical University
Locations (1):
- Beijing Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 2025.5-
Access Criteria: via reasonable email requests

REFERENCES:
- [Background] Bosset JF, Calais G, Mineur L, Maingon P, Radosevic-Jelic L, Daban A, Bardet E, Beny A, Briffaux A, Collette L. Enhanced tumorocidal effect of chemotherapy with preoperative radiotherapy for rectal cancer: preliminary results--EORTC 22921. J Clin Oncol. 2005 Aug 20;23(24):5620-7. doi: 10.1200/JCO.2005.02.113. Epub 2005 Jul 11. PMID 16009958
- [Background] Gerard JP, Conroy T, Bonnetain F, Bouche O, Chapet O, Closon-Dejardin MT, Untereiner M, Leduc B, Francois E, Maurel J, Seitz JF, Buecher B, Mackiewicz R, Ducreux M, Bedenne L. Preoperative radiotherapy with or without concurrent fluorouracil and leucovorin in T3-4 rectal cancers: results of FFCD 9203. J Clin Oncol. 2006 Oct 1;24(28):4620-5. doi: 10.1200/JCO.2006.06.7629. PMID 17008704
- [Background] Hata T, Takahashi H, Sakai D, Haraguchi N, Nishimura J, Kudo T, Chu M, Takemasa I, Taroh S, Mizushima T, Doki Y, Mori M. Neoadjuvant CapeOx therapy followed by sphincter-preserving surgery for lower rectal cancer. Surg Today. 2017 Nov;47(11):1372-1377. doi: 10.1007/s00595-017-1527-5. Epub 2017 May 4. PMID 28474202
- [Background] Shamseddine A, Zeidan YH, El Husseini Z, Kreidieh M, Al Darazi M, Turfa R, Kattan J, Khalifeh I, Mukherji D, Temraz S, Alqasem K, Amarin R, Al Awabdeh T, Deeba S, Jamali F, Mohamad I, Elkhaldi M, Daoud F, Al Masri M, Dabous A, Hushki A, Jaber O, Charafeddine M, Geara F. Efficacy and safety-in analysis of short-course radiation followed by mFOLFOX-6 plus avelumab for locally advanced rectal adenocarcinoma. Radiat Oncol. 2020 Oct 7;15(1):233. doi: 10.1186/s13014-020-01673-6. PMID 33028346
- [Background] Shen Z, Bu Z, Li A, Lu J, Zhu L, Chong CS, Gao Z, Jiang K, Wang S, Li F, Xiao Y, Ji J, Ye Y. Multicenter study of surgical and oncologic outcomes of extra-levator versus conventional abdominoperineal excision for lower rectal cancer. Eur J Surg Oncol. 2020 Jan;46(1):115-122. doi: 10.1016/j.ejso.2019.08.017. Epub 2019 Aug 21. PMID 31471089
- [Background] Wu F, Zhou C, Wu B, Zhang X, Wang K, Wang J, Xiao L, Wang G. Adding Adjuvants to Fluoropyrimidine-based Neoadjuvant Chemoradiotherapy for Locally Advanced Rectal Cancer: An Option Worthy of Serious Consideration. J Cancer. 2021 Jan 1;12(2):417-427. doi: 10.7150/jca.48337. eCollection 2021. PMID 33391438
- [Background] Chen W, Zheng R, Baade PD, Zhang S, Zeng H, Bray F, Jemal A, Yu XQ, He J. Cancer statistics in China, 2015. CA Cancer J Clin. 2016 Mar-Apr;66(2):115-32. doi: 10.3322/caac.21338. Epub 2016 Jan 25. PMID 26808342
- [Background] Chen WZ, Chen XD, Ma LL, Zhang FM, Lin J, Zhuang CL, Yu Z, Chen XL, Chen XX. Impact of Visceral Obesity and Sarcopenia on Short-Term Outcomes After Colorectal Cancer Surgery. Dig Dis Sci. 2018 Jun;63(6):1620-1630. doi: 10.1007/s10620-018-5019-2. Epub 2018 Mar 16. PMID 29549473
- [Background] Lawler M, Alsina D, Adams RA, Anderson AS, Brown G, Fearnhead NS, Fenwick SW, Halloran SP, Hochhauser D, Hull MA, Koelzer VH, McNair AGK, Monahan KJ, Nathke I, Norton C, Novelli MR, Steele RJC, Thomas AL, Wilde LM, Wilson RH, Tomlinson I; Bowel Cancer UK Critical Research Gaps in Colorectal Cancer Initiative. Critical research gaps and recommendations to inform research prioritisation for more effective prevention and improved outcomes in colorectal cancer. Gut. 2018 Jan;67(1):179-193. doi: 10.1136/gutjnl-2017-315333. PMID 29233930
- [Background] Sung JJY, Chiu HM, Jung KW, Jun JK, Sekiguchi M, Matsuda T, Kyaw MH. Increasing Trend in Young-Onset Colorectal Cancer in Asia: More Cancers in Men and More Rectal Cancers. Am J Gastroenterol. 2019 Feb;114(2):322-329. doi: 10.14309/ajg.0000000000000133. PMID 30694865
- [Background] Cao Y, Li W, Wang Z, Pang H. Potential and unsolved problems of anti-PD-1/PD-L1 therapy combined with radiotherapy. Tumori. 2021 Aug;107(4):282-291. doi: 10.1177/0300891620940382. Epub 2020 Jul 31. PMID 32734832
- [Derived] Gao J, Zhang X, Yang Z, Zhang J, Bai Z, Deng W, Chen G, Xu R, Wei Q, Liu Y, Han J, Li A, Liu G, Sun Y, Kong D, Yao H, Zhang Z. Interim result of phase II, prospective, single-arm trial of long-course chemoradiotherapy combined with concurrent tislelizumab in locally advanced rectal cancer. Front Oncol. 2023 Feb 2;13:1057947. doi: 10.3389/fonc.2023.1057947. eCollection 2023. PMID 36816939
- [Derived] Yang Z, Zhang X, Zhang J, Gao J, Bai Z, Deng W, Chen G, An Y, Liu Y, Wei Q, Han J, Li A, Liu G, Sun Y, Kong D, Yao H, Zhang Z. Rationale and design of a prospective, multicenter, phase II clinical trial of safety and efficacy evaluation of long course neoadjuvant chemoradiotherapy plus tislelizumab followed by total mesorectal excision for locally advanced rectal cancer (NCRT-PD1-LARC trial). BMC Cancer. 2022 Apr 27;22(1):462. doi: 10.1186/s12885-022-09554-9. PMID 35477432